CLINICAL TRIAL: NCT03901976
Title: ZeroFall - Reliability Testing of Optical Sensor to Detect Bed Exit for Patients in Hospital
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough resources in place; COVID-19 pandemic impedes working on the project and travelling within the EU
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: YGB-PH-CS-BD-2018-02-18
Record Dates: First submitted 2019-03-28; First posted 2019-04-03 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Delirium of Mixed Origin
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Intervention Model Description: The study has several distinct phases:
  * Silent Phase: The devices run in the background, activity is blinded for clinicians, settings are optimized by the research team.
  * Run-In Phase: Bed exit notifications are turned on, notifications will be configurable for acceptability by clinical teams. Data extraction and data evaluation will be tested.
  * Phase I: Data collection of bed exit data of sensors as well as data related to falls
  * Phase II: Data collection of bed exit data with optimization of predictive algorithms
  * Phase III: Data collection for validation using predictive data for early notification
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bed Exit Detection On (Other): prevention of fall by a true bed exit detection
  Interventions: Device: bed exit detection

INTERVENTIONS:
Device: bed exit detection — bed exit detection to avoid patients fall

SUMMARY:
Falls are one of the most common NHS adverse events. With an increasing number of frail elderly patients being admitted this risk is likely to increase. In order to be able to assist patients with bed exit in a timely manner monitoring might be of help. In ZeroFall we will test the reliability of monitoring devices to notify care givers if a patient is attempting to exit the bed.

DETAILED DESCRIPTION:
In ZeroFall we intend to observe patients on risk of fall with two different devices during their hospital stay: The information from a no-touch optical sensing device that analyses movement and an under the mattress sensor that has already been used in a previous study at Bangor. Both are compatible with an existing monitoring system by Philips Healthcare and CE marked.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with risk of fall more than 24 hours on the ward

Exclusion Criteria:

Patients with predominantly palliative needs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Number of true bed exit detections vs number of false bed exit detections | 12-15 months
  A reference device and two observers will classify if a bed exit was true

CONTACTS AND LOCATIONS:
Overall Officials: Christian P Subbe, MD, Principal Investigator — Ysbyty Gwynedd Hospital
Locations (1):
- Ysbyty Gwynedd, Bangor, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No